CLINICAL TRIAL: NCT03177889
Title: Efficacy and Safety of Lung Dispersing, Turbid Descending and Gut Clearing Decoction on Clinically Stable Bronchiectasis (LUNG-CLEAR): A Multicenter, Randomized, Cross-over Trial
Brief Title: Lung Dispersing, Turbid Descending and Gut Clearing Decoction for Bronchiectasis
Acronym: LUNG-CLEAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Weijie Guan, associate professor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GWJ-TCM-2017
Record Dates: First submitted 2017-06-04; First posted 2017-06-06 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Bronchiectasis Adult; Traditional Chinese Medicine; Quality of Life; Exacerbation
MeSH Terms: interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual treatment (Sham Comparator): oral mucolytics [ambroxol 30mg tid, or N-acetylcysteine 0.2g tid, serrapeptase 10mg tid, or carbocisteine 500mg tid]
  Interventions: Combination Product: Traditional Chinese Medicine (TCM)
- TCM treatment (Active Comparator): Traditional Chinese Medicine plus oral mucolytics (described above);
  Agastache rugosus 5g, Scutellaria baicalensis 10g, Radix Puerariae 10g, Acorus tatarinowii schott 10g, Fructus Liquidambaris 5g, gypsum 15 g, Rheum officinale 5 g, Folium sennae 5 g, Codonopsis pilosula 10g, Radix Salviae Miltiorrhizae 10g, Lignum millettiae 10 g, Liquiritia glycyrrhiza 10 g
  Interventions: Combination Product: Traditional Chinese Medicine (TCM)

INTERVENTIONS:
Combination Product: Traditional Chinese Medicine (TCM) — Traditional Chinese Medicine plus oral mucolytics [ambroxol 30mg tid, or N-acetylcysteine 0.2g tid, serrapeptase 10mg tid, or carbocisteine 500mg tid];
  Agastache rugosus 5g, Scutellaria baicalensis 10g, Radix Puerariae 10g, Acorus tatarinowii schott 10g, Fructus Liquidambaris 5g, gypsum 15 g, Rheum officinale 5 g, Folium sennae 5 g, Codonopsis pilosula 10g, Radix Salviae Miltiorrhizae 10g, Lignum millettiae 10 g, Liquiritia glycyrrhiza 10 g
  Optional formulae: bile arisaema 15g, polygala tenuifolia 15g, Mangnolia officinalis 10g, Fructus aurantii immaturus 10g; Magnetite 15-30g and reddle15-30g
  Other Names: TCM

SUMMARY:
Bronchiectasis is a chronic airway disease which confers significant healthcare burden, with limited therapeutic approaches. From the perspective of traditional Chinese medicine, congenital insufficiency of the lung, spleen and kidney, when coupled with external injury or mood impairment, may collectively contribute to bronchiectasis pathogenesis due to heat trapping in the phlems, congestion of wind evils and stagnation of blood. Here, the investigators will explore the Lung Dispersing, Turbid Descending and Gut Clearing Decoction (LTGD) which targets at expelling the wind evil in patients with bronchiectasis. The investigators sought to conduct a multicenter, randomized cross-over trial which investigates the efficacy and safety of LTGD on clinically stable bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic airway disease which confers significant healthcare burden, with limited therapeutic approaches. From the perspective of traditional Chinese medicine, congenital insufficiency of the lung, spleen and kidney, when coupled with external injury or mood impairment, may collectively contribute to bronchiectasis pathogenesis due to heat trapping in the phlems, congestion of wind evils and stagnation of blood. Symptomatic treatment may be effective and safe for ameliorating respiratory symptoms and hindering disease progression of bronchiectasis. Here, the investigators have explored the Lung Dispersing, Turbid Descending and Gut Clearing Decoction (LTGD) which targets at expelling the wind evil in patients with bronchiectasis. The investigators sought to conduct a multicenter, randomized cross-over trial which investigates the efficacy and safety of LTGD on clinically stable bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 75 years;
* remained clinically stable (respiratory symptoms and lung function parameters not exceeding normal daily variations) for 4 consecutive weeks;
* no acute upper respiratory tract infections within 4 weeks;
* 1 or more BEs within the previous 2 years

Exclusion Criteria:

* Other unstable concomitant systemic illnesses (i.e. coronary heart disease, recent cerebral stroke, severe uncontrolled hypertension, active gastric or duodenal ulcer, uncontrolled diabetes, malignancy, hepatic or renal dysfunction);
* Concomitant asthma, allergic bronchopulmonary aspergillosis, or active tuberculosis;
* Concomitant chronic obstructive pulmonary disease as the predominant diagnosis;
* Treatment with inhaled, oral or systemic antibiotics within 4 weeks;
* Type 2 respiratory failure needing oxygen therapy or non-invasive mechanical ventilation;
* Females during lactation or pregnancy;
* Poor understanding or failure to properly operate the instrument;
* Participation in other clinical trials within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Bronchiectasis Health Questionnaire scores at month 6 compared with baseline | 6 months
  Changes in Bronchiectasis Health Questionnaire scores at month 6 compared with baseline

SECONDARY OUTCOMES:
the frequency of bronchiectasis exacerbation | 6 months
  the frequency of bronchiectasis exacerbation
the time to the first bronchiectasis exacerbation | 6 months
  the time to the first bronchiectasis exacerbation
changes in forced expiratory volume in one second at month 6 compared with baseline | 6 months
  changes in forced expiratory volume in one second at month 6 compared with baseline
24-hour sputum volume at month 6 compared with baseline | 6 months
  24-hour sputum volume at month 6 compared with baseline
changes in sputum purulence score at month 6 compared with baseline | 6 months
  changes in sputum purulence score at month 6 compared with baseline
the proportion of patients isolated with Pseudomonas aeruginosa at month 6 compared with baseline | 6 months
  the proportion of patients isolated with Pseudomonas aeruginosa at month 6 compared with baseline

OTHER OUTCOMES:
changes in sputum hydrogen peroxide level at month 6 compared with baseline | 6 months
  changes in sputum hydrogen peroxide level at month 6 compared with baseline
changes in sputum catalase activity at month 6 compared with baseline | 6 months
  changes in sputum catalase activity at month 6 compared with baseline
changes in sputum total antioxidant capacity at month 6 compared with baseline | 6 months
  changes in sputum total antioxidant capacity at month 6 compared with baseline
changes in airway resistance measured at 5 Hz at month 6 compared with baseline | 6 months
  changes in airway resistance measured at 5 Hz at month 6 compared with baseline
changes in Quality-of-life-bronchiectasis questionnaire score at month 6 compared with baseline | 6 months
  changes in Quality-of-life-bronchiectasis questionnaire score at month 6 compared with baseline
changes in sputum microbiota composition at month 6 compared with baseline | 6 months
  changes in sputum microbiota composition at month 6 compared with baseline
Changes in AX at month 6 compared with baseline | 6 months
  Changes in AX at month 6 compared with baseline
Changes in sputum superoxide dismutase activity at month 6 compared with baseline | 6 months
  Changes in sputum superoxide dismutase activity at month 6 compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wei-jie Guan, MD, Study Chair — First Affiliated Hospital of Guangzhou Medical University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Pasteur MC, Bilton D, Hill AT; British Thoracic Society Non-CF Bronchiectasis Guideline Group. British Thoracic Society guideline for non-CF bronchiectasis. Thorax. 2010 Jul;65(7):577. doi: 10.1136/thx.2010.142778. No abstract available. PMID 20627912
- [Background] Loukides S, Horvath I, Wodehouse T, Cole PJ, Barnes PJ. Elevated levels of expired breath hydrogen peroxide in bronchiectasis. Am J Respir Crit Care Med. 1998 Sep;158(3):991-4. doi: 10.1164/ajrccm.158.3.9710031. PMID 9731036
- [Background] Horvath I, Loukides S, Wodehouse T, Kharitonov SA, Cole PJ, Barnes PJ. Increased levels of exhaled carbon monoxide in bronchiectasis: a new marker of oxidative stress. Thorax. 1998 Oct;53(10):867-70. doi: 10.1136/thx.53.10.867. PMID 10193374
- [Background] Tsang KW, Chan K, Ho P, Zheng L, Ooi GC, Ho JC, Lam W. Sputum elastase in steady-state bronchiectasis. Chest. 2000 Feb;117(2):420-6. doi: 10.1378/chest.117.2.420. PMID 10669685
- [Background] Quittner AL, O'Donnell AE, Salathe MA, Lewis SA, Li X, Montgomery AB, O'Riordan TG, Barker AF. Quality of Life Questionnaire-Bronchiectasis: final psychometric analyses and determination of minimal important difference scores. Thorax. 2015 Jan;70(1):12-20. doi: 10.1136/thoraxjnl-2014-205918. Epub 2014 Oct 16. PMID 25323621
- [Background] Spinou A, Siegert RJ, Guan WJ, Patel AS, Gosker HR, Lee KK, Elston C, Loebinger MR, Wilson R, Garrod R, Birring SS. The development and validation of the Bronchiectasis Health Questionnaire. Eur Respir J. 2017 May 11;49(5):1601532. doi: 10.1183/13993003.01532-2016. Print 2017 May. PMID 28495688
- [Background] Zheng J, Zhong N. Normative values of pulmonary function testing in Chinese adults. Chin Med J (Engl). 2002 Jan;115(1):50-4. PMID 11930658
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Sputum bacteriology in steady-state bronchiectasis in Guangzhou, China. Int J Tuberc Lung Dis. 2015 May;19(5):610-9. doi: 10.5588/ijtld.14.0613. PMID 25868032
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Gu YY, Liu GH, Li HM, Chen RC, Zhong NS. Sputum matrix metalloproteinase-8 and -9 and tissue inhibitor of metalloproteinase-1 in bronchiectasis: clinical correlates and prognostic implications. Respirology. 2015 Oct;20(7):1073-81. doi: 10.1111/resp.12582. Epub 2015 Jun 30. PMID 26122009
- [Result] Zhang ZM, Ren PH, Wu ZJ, Zhang DP, Xie WJ. Personalized alternative therapy of intractable bronchiectasis-induced hemoptysis in a patient: syndrome differentiation and treatment according to individual physique category. J Thorac Dis. 2013 Jun;5(3):E115-7. doi: 10.3978/j.issn.2072-1439.2013.06.26. No abstract available. PMID 23825784
- [Result] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Impulse oscillometry in adults with bronchiectasis. Ann Am Thorac Soc. 2015 May;12(5):657-65. doi: 10.1513/AnnalsATS.201406-280OC. PMID 25654540